CLINICAL TRIAL: NCT05111860
Title: Efficacy and Safety of Neoadjuvant Bevacizumab + Chemotherapy Combined With Short-course Radiotherapy for RAS Mutant-type Locally Advanced Rectal Cancer
Brief Title: Neoadjuvant Bevacizumab + Chemotherapy Combined With Short-course Radiotherapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MISC-Bev-SCRT
Record Dates: First submitted 2021-10-25; First posted 2021-11-08 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Neoadjuvant Treatment; Rectal Cancer; Bevacizumab; Radiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental)
  Interventions: Drug: Bevacizumab+mFOLFOX6

INTERVENTIONS:
Drug: Bevacizumab+mFOLFOX6 — Bevacizumab 5mg/kg d1 Oxaliplatin 85mg/m2 d1 Calcium Folinate 400mg/m2 d1 5-fluorouridine 400mg/m2 d1 5-fluorouridine 2400mg/m2 46h q2w, 6 cycles

SUMMARY:
Prospectively Investigate the effectiveness and safety of neoadjuvant Bevacizumab + chemotherapy (mFOLFOX6) combined with short-course radiotherapy (25Gy/5Fx) for RAS mutant-type locally advanced rectal cancer

ELIGIBILITY:
Inclusion Criteria:

1. A biopsy proven histological diagnosis of rectal adenocarcinoma；
2. An ARMS-PCR proven KRAS, NRAS mutation, excluding BRAF mutation or microsatellite instablility-High;
3. No intestinal obstruction, distant metastasis was excluded by CT, MRI or PET / CT;
4. MRI proven T3c-T4, CRM positive, N2, extramural vascular invasion positive or lateral lymph node positive of locally advanced rectal cancer;
5. Age between 18-75 years;
6. ECOG (Eastern US Cooperative Oncology Group) score: 0-1;
7. Has sufficient organ function:

   * Hemopoietic function: hemoglobin ≥ 90 g / L, platelet ≥ 80 g / L × 109 / L,
   * neutrophils ≥ 1.5 × 109/L
   * Liver function: ALT and AST < 2.5 × ULN;
   * Renal function: serum creatinine < 1.5 ULN;
8. Willing to participate and informed consent signed；

Exclusion Criteria:

1. An ARMS-PCR proven RAS wild type, BRAF mutation and microsatellite instablility-High;
2. Patients having undergone chemotherapy, radiotherapy or surgery for colorectal cancer;
3. Patients with other uncontrolled malignant tumors (except early-stage basal cell carcinoma or cervical carcinoma in situ) ;
4. Female patients who are pregnant or breastfeeding;
5. Patients with severe heart, liver, or kidney, or neurological or psychiatric disease;
6. Patients with active infection;
7. Poor overall health status, ECOG ≥ 2;
8. Patients with concomitant diseases that seriously endanger the safety of patients or affect the completion of the study in the judgment of the investigator;
9. Known hypersensitivity reactions to any investigational drugs;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Peri-operative complications | From the start of treatment to 3 months after surgery
  Complications occurring in the perioperative period

SECONDARY OUTCOMES:
Pathological response rate | 2 weeks after surgery
  Tumor Regression Grade 0-1
Pathological complete response rate | 2 weeks after surgery
  Refers to the pathological examination of primary tumors and lymph node surgical specimens without residual infiltrating tumor cells (ypT0N0, TRG 0)
2-year local control rate | 2 years
  Refers to the probability of not finding local recurrence of tumor within 2 years，including anastomotic recurrence confirmed by pathological biopsy, pelvic tumor recurrence confirmed by imaging examination, or suspected pelvic recurrence with CEA exceeding the normal upper limit.
2-year metastasis-free rate | 2 years
  Refers to the probability of no distant metastasis within 2 years
Overall survival | 2 years
  Refers to the time from the start of treatment to death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China